CLINICAL TRIAL: NCT03284827
Title: a Multicenter, Randomized, Open-label, Active-treatment, Controlled Trial to Compare the Efficacy of NOAC With Edoxaban vs. Dual Antiplatelet Therapy (DAPT) for Prevention of Leaflet Thrombosis (Documented by Cardiac CT Imaging) and Cerebral Embolization (Documented With Brain DW-MRI Imaging) in Patients Without an Absolute Indication for Chronic OAC After Successful TAVR
Brief Title: Anticoagulant Versus Dual Antiplatelet Therapy for Preventing Leaflet Thrombosis and Cerebral Embolization After Transcatheter Aortic Valve Replacement
Acronym: ADAPT-TAVR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMCCV 2017-08
Record Dates: First submitted 2017-09-12; First posted 2017-09-15 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Aortic Valve Stenosis
Keywords: edoxaban; dual antiplatelet therapy; cerebral embolization; leaflet thrombosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOAC (Experimental): 60 mg once daily
  Interventions: Drug: NOAC
- DAPT (Active Comparator): clopidogrel (75 mg OD) plus acetylsalicylic acid (ASA, 75-100 mg OD)
  Interventions: Drug: DAPT

INTERVENTIONS:
Drug: NOAC — edoxaban (60 mg once daily [OD]) for at least 6 months
  Arms: NOAC
Drug: DAPT — clopidogrel (75 mg OD) plus acetylsalicylic acid (ASA, 75-100 mg OD) for at least 6 months
  Arms: DAPT

SUMMARY:
This trial is to compare the efficacy of NOAC(Novel Oral Anticoagulants) with edoxaban vs. dual antiplatelet therapy (DAPT) for prevention of leaflet thrombosis (documented by cardiac CT imaging) and cerebral embolization (documented with brainDiffusion-weighted (DW) magnetic resonance (MR) imaging) in patients without an absolute indication for chronic oral anticoagulation (OAC) after successful transcatheter aortic valve replacement(TAVR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age or older with successful TAVR procedure

   * either native valve or valve-in-valve with any approved/marketed device
   * A successful TAVR is defined as device success according to the VARC-2 criteria:

     1. correct positioning of a single prosthetic heart valve into the proper anatomical location AND
     2. Intended performance of the prosthetic heart valve (no prosthesis- patient mismatch* and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, no moderate or severe prosthetic valve regurgitation AND
     3. absence of periprocedural complications (any type of stroke, life-threatening bleeding, acute coronary artery obstruction requiring intervention, major vascular complication requiring intervention, unresolved acute valve thrombosis, or any requirement of a repeat procedure.
2. Patients who voluntarily participated in the written agreement

Exclusion Criteria:

1. Any atrial fibrillation with an indication for chronic OAC.
2. An ongoing indication for OAC or any other indication for continued treatment with any OAC
3. Any ongoing indication for DAPT (recent acute coronary syndrome or PCI within 12 months)
4. Planned coronary or vascular intervention or major surgery
5. Clinically significant bleeding patients
6. The risk of bleeding increased due to the following reasons at the time of TAVR procedure, i. history of gastrointestinal ulcers within 1 month ii. Malignant tumor with high risk of bleeding iii. Brain or spinal cord injury within 1 month iv. History of intracranial or intracerebral hemorrhage within 12 months v. Esophageal varices vi. Arteriovenous malformation vii. Vascular aneurysms viii. Spinal cord vascular abnormalities or intracerebral vascular abnormalities ix. Active bleeding x. Hemoglobin level <7.0 g/dL or platelet count ≤ 50,000 / mm3 xi. History of major surgery within 1 month
7. Clinically overt stroke within the last 3 months
8. Moderate and severe hepatic impairment, and any hepatic disease associated with coagulopathy
9. Severe renal impairment (CrCl by Cockcroft-Gault equation<15 mL/min per 1.73 m2), chronic dialysis, or post-TAVR unresolved acute kidney injury
10. Terminal illness with life expectancy <6 months
11. Hypersensitivity to the main component or constituents of Edoxaban
12. Severe hypertensive patient
13. Patient who received prosthetic heart valve replacement for which anticoagulant therapy is essential
14. Moderate to severe mitral stenosis
15. Pulmonary embolism requiring thrombolysis or pulmonary embolectomy
16. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
17. Pregnancy test results are positive (all pregnant women should undergo urinary human chorionic gonadotropin (hCG) testing within 7 days prior to screening and / or randomization) or during pregnancy or lactation
18. Genetic problem with galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
19. History of hypersensitivity to Edoxaban, Aspirin or clopidogrel
20. Current or history of Aspirin- or NSAIDs-induced asthma
21. Hemophilia
22. Patients who are using Methotrexate at doses of 15mg or more per week
23. Patients who have unsuitable condition to undergo Brain MRI(Magnetic resonance imaging) and/or Cardiac CT(computed tomography) (e.g., tremor from Parkinson's disease). This is at the discretion of investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
an incidence of leaflet thrombosis | 6-month
  an incidence of leaflet thrombosis on four-dimensional, volume-rendered cardiac CT imaging

SECONDARY OUTCOMES:
Death | 6-month
  all-cause, cardiovascular, or non-cardiovascular mortality
Myocardial infarction | 6-month
Stroke or transient ischemic attack | 6-month
  disabling or non-disabling
Bleeding event | 6-month
  life-threatening or disabling, major bleeding, or minor bleeding according to VARC(The Valve Academic Research Consortium)-2 definition
The change of Echocardiographic parameter | 6-month
  the mean transaortic valve pressure gradient and velocity time integral ratio at baseline and 6-month follow-up
New lesion volume on MRI scans | 6-month
The change of neurological and neurocognitive function | 6-month
  according to NeuroARC(Neuro Academic Research Consortium) definition
the number of new lesions on brain DW-MRI scans | 6-month
  the number of new lesions on brain DW-MRI scans at 6 months relative to immediate post-TAVR

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, Principal Investigator — Cardiology, Asan Medical Center Heart Institute
Locations (5):
- Queen Mary Hospital, Hong Kong, Hong Kong
- South Korea (2):
  - Asan Medical Center, Seoul, Songpa-gu
  - Bundang CHA Hospital, Seongnam
- Taiwan (2):
  - Cheng Hsin General Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi Y, Ahn JM, Kang DY, Kim HJ, Kim H, Lee J, Kim M, Park J, Kim KW, Koo HJ, Yang DH, Jung SC, Kim B, Anthony Wong YT, Simon Lam CC, Yin WH, Wei J, Lee YT, Kao HL, Lin MS, Ko TY, Kim WJ, Kang SH, Lee SA, Kim DH, Lee JH, Park SJ, Park DW; ADAPT-TAVR Investigators. Frequency, Predictors, and Clinical Impact of Valvular and Perivalvular Thrombus After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2023 Dec 25;16(24):2967-2981. doi: 10.1016/j.jcin.2023.10.024. PMID 38151311
- [Derived] Jang MH, Ahn JM, Kang DY, Kim KW, Koo HJ, Yang DH, Jung SC, Kim B, Wong YTA, Lam CCS, Yin WH, Wei J, Lee YT, Kao HL, Lin MS, Ko TY, Kim WJ, Kang SH, Ko E, Lee SA, Kim DH, Kim H, Choi Y, Lee J, Park SJ, Park DW. Impact of leaflet thrombosis on valve haemodynamic status after transcatheter aortic valve replacement. Heart. 2023 Dec 20;110(2):140-147. doi: 10.1136/heartjnl-2023-322946. PMID 37586823
- [Derived] Park DW, Ahn JM, Kang DY, Kim KW, Koo HJ, Yang DH, Jung SC, Kim B, Wong YTA, Lam CCS, Yin WH, Wei J, Lee YT, Kao HL, Lin MS, Ko TY, Kim WJ, Kang SH, Yun SC, Lee SA, Ko E, Park H, Kim DH, Kang JW, Lee JH, Park SJ; ADAPT-TAVR Investigators. Edoxaban Versus Dual Antiplatelet Therapy for Leaflet Thrombosis and Cerebral Thromboembolism After TAVR: The ADAPT-TAVR Randomized Clinical Trial. Circulation. 2022 Aug 9;146(6):466-479. doi: 10.1161/CIRCULATIONAHA.122.059512. Epub 2022 Apr 4. PMID 35373583
- [Derived] Park H, Kang DY, Ahn JM, Kim KW, Wong AYT, Lam SCC, Yin WH, Wei J, Lee YT, Kao HL, Lin MS, Ko TY, Kim WJ, Kang SH, Ko E, Kim DH, Koo HJ, Yang DH, Kang JW, Jung SC, Lee JH, Yun SC, Park SJ, Park DW. Rationale and design of the ADAPT-TAVR trial: a randomised comparison of edoxaban and dual antiplatelet therapy for prevention of leaflet thrombosis and cerebral embolisation after transcatheter aortic valve replacement. BMJ Open. 2021 Jan 5;11(1):e042587. doi: 10.1136/bmjopen-2020-042587. PMID 33402409